CLINICAL TRIAL: NCT00853840
Title: A Randomized, Single-Blinded, Placebo-Controlled Two-Way Crossover Study To Investigate The Hemodynamic Effects Of Single Dose Vardenafil In Subjects Receiving Maraviroc
Brief Title: Study To Investigate The Hemodynamic Effects Of Single Dose Vardenafil In Subjects Receiving Maraviroc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A4001074
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: AIDS
Keywords: pharmacodynamics. maraviroc, vardenafil, blood pressure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. (Experimental): Maraviroc + Vardenafil
  Interventions: Drug: Maraviroc; Drug: Vardenafil
- 2. (Placebo Comparator): Maraviroc + Placebo
  Interventions: Drug: Maraviroc; Drug: Placebo

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 300 mg twice daily for 3 - 4 days plus a single oral dose of Vardenafil 20 mg.
  Other Names: Celsentri, Selzentry
  Arms: 1.
Drug: Vardenafil — Maraviroc 300 mg twice daily for 3 - 4 days plus a single oral dose of Vardenafil 20 mg.
  Arms: 1.
Drug: Maraviroc — Maraviroc 300 mg twice daily for 3 - 4 days plus a single oral dose of Placebo.
  Other Names: Selzentry, Celsentri
  Arms: 2.
Drug: Placebo — Maraviroc 300 mg twice daily for 3 - 4 days plus a single oral dose of Placebo.
  Arms: 2.

SUMMARY:
The objective of this study was to estimate the effects of a single dose of vardenafil on the blood pressure (BP) in subjects receiving maraviroc (MVC) (dosed to steady-state) and to assess the safety and tolerability of MVC in subjects receiving a single dose of vardenafil.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects. no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram and clinical laboratory tests.
* Body mass index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Subjects with a supine systolic BP of greater than 140 mm Hg, or a supine diastolic BP of greater than 90 mm Hg, either at Screening or at the predose measurements.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001074&StudyName=Study%20To%20Investigate%20The%20Hemodynamic%20Effects%20Of%20Single%20Dose%20Vardenafil%20In%20Subjects%20Receiving%20Maraviroc

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects received 3 to 4 days of maraviroc 300 mg twice daily (BID) before receiving single oral doses of either vardenafil 20 mg (Treatment A) or placebo (Treatment B).
Groups:
- Vardenafil + Maraviroc: On Days 1 through 3 during Period 1, and Days 1 through 2 during Period 2, a maraviroc 300 mg tablet was taken orally BID to achieve steady state. On Day 4 of Period 1, and Day 3 of Period 2, a single dose of vardenafil 20 mg tablet was administered orally 1 hour post maraviroc dosing.
- Non-matching Placebo + Maraviroc: On Days 1 through 3 during Period 1, and Days 1 through 2 during Period 2, a maraviroc 300 mg tablet was taken orally BID to achieve steady state. On Day 4 of Period 1, and Day 3 of Period 2, a single dose of a non-matching placebo tablet was administered orally 1 hour post maraviroc dosing.
Period: Period 1
Arm/Group | Vardenafil + Maraviroc | Non-matching Placebo + Maraviroc
Started | 9 | 9
Maraviroc (Days 1 - 4) | 9 | 9
Vardenafil or Placebo (Day 4) | 9 (Administered 1 hour post Maraviroc dosing) | 9 (Administered 1 hour post Maraviroc dosing)
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Vardenafil + Maraviroc | Non-matching Placebo + Maraviroc
Started | 9 | 9
Maraviroc (Days 1 - 3) | 9 | 9
Vardenafil or Placebo (Day 3) | 9 (Administered 1 hour post Maraviroc dosing) | 9 (Administered 1 hour post Maraviroc dosing)
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: In this 2-way crossover study, in Period 1, all 18 subjects were randomized to receive a single dose of either vardenafil 20 mg (Treatment A) or placebo (Treatment B), subsequent to treatment with 3 to 4 days of maraviroc 300 mg BID. All subjects were then crossed over to receive the second treatment in Period 2.
Arm/Group | All Subjects
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 34.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Standing and Supine Systolic and Diastolic Blood Pressure (BP)
Description: Supine BP was taken after subjects rested for 5 minutes supine. Subjects then sat for 2 minutes and stood for 2 minutes then standing BP taken. Duplicate supine and standing BP measurements were taken per the protocol. The average of the duplicate measurements was calculated prior to data analysis.
Time Frame: 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours post Vardenafil or Placebo dose
Population: The vital sign analysis population was defined as all enrolled subjects who received at least 1 dose of study medication and had at least 1 vital sign parameter in at least 1 treatment period.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Maraviroc + Vardenafil (Treatment A): On Days 1 through 3 during Period 1, and Days 1 through 2 during Period 2, a maraviroc 300 mg tablet was taken orally BID to achieve steady state. On Day 4 of Period 1, and Day 3 of Period 2, a single dose of vardenafil 20 mg tablet was administered orally 1 hour post maraviroc dosing.
- Maraviroc + Placebo (Treatment B): On Days 1 through 3 during Period 1, and Days 1 through 2 during Period 2, a maraviroc 300 mg tablet was taken orally BID to achieve steady state. On Day 4 of Period 1, and Day 3 of Period 2, a single dose of a non-matching placebo tablet was administered orally 1 hour post maraviroc dosing.
Arm/Group | Maraviroc + Vardenafil (Treatment A) | Maraviroc + Placebo (Treatment B)
Number analyzed (Participants) | 18 | 18
mm Hg
  Supine Systolic BP: 1.5 hour post Maraviroc dose | 118.36 (1.1523) | 119.47 (1.1523)
  Supine Diastolic BP: 1.5 hour post Maraviroc dose | 68.06 (0.7184) | 69.99 (0.7184)
  Supine Systolic BP: 2 hour post Maraviroc dose | 113.45 (1.1523) | 118.44 (1.1523)
  Supine Diastolic BP: 2 hour post Maraviroc dose | 66.31 (0.7184) | 69.27 (0.7184)
  Supine Systolic BP: 2.5 hour post Maraviroc dose | 114.67 (1.1523) | 119.55 (1.1523)
  Supine Diastolic BP: 2.5 hour post Maraviroc dose | 66.98 (0.7184) | 70.80 (0.7184)
  Supine Systolic BP: 3 hour post Maraviroc dose | 114.11 (1.1523) | 116.16 (1.1523)
  Supine Diastolic BP: 3 hour post Maraviroc dose | 67.28 (0.7184) | 69.05 (0.7184)
  Supine Systolic BP: 4 hour post Maraviroc dose | 115.89 (1.1523) | 117.97 (1.1523)
  Supine Diastolic BP: 4 hour post Maraviroc dose | 68.37 (0.7184) | 69.24 (0.7184)
  Supine Systolic BP: 6 hour post Maraviroc dose | 116.45 (1.1523) | 118.75 (1.1523)
  Supine Diastolic BP: 6 hour post Maraviroc dose | 65.67 (0.7184) | 66.52 (0.7184)
  Supine Systolic BP: 8 hour post Maraviroc dose | 116.61 (1.1523) | 120.83 (1.1523)
  Supine Diastolic BP: 8 hour post Maraviroc dose | 66.34 (0.7184) | 68.85 (0.7184)
  Supine Systolic BP: 12 hour post Maraviroc dose | 122.81 (1.1523) | 124.75 (1.1523)
  Supine Diastolic BP: 12 hour post Maraviroc dose | 67.95 (0.7184) | 70.27 (0.7184)
  Standing Systolic BP: 1.5 hour post Maraviroc dose | 120.82 (1.6525) | 125.18 (1.6525)
  Standing Diastolic BP 1.5 hour post Maraviroc dose | 74.81 (1.0102) | 78.74 (1.0102)
  Standing Systolic BP: 2 hour post Maraviroc dose | 118.49 (1.6525) | 125.40 (1.6525)
  Standing Diastolic BP: 2 hour post Maraviroc dose | 74.90 (1.0102) | 80.69 (1.0102)
  Standing Systolic BP: 2.5 hour post Maraviroc dose | 115.52 (1.6525) | 121.32 (1.6525)
  Standing Diastolic BP 2.5 hour post Maraviroc dose | 72.29 (1.0102) | 78.94 (1.0102)
  Standing Systolic BP: 3 hour post Maraviroc dose | 117.10 (1.6525) | 121.37 (1.6525)
  Standing Diastolic BP: 3 hour post Maraviroc dose | 73.73 (1.0102) | 77.38 (1.0102)
  Standing Systolic BP: 4 hour post Maraviroc dose | 119.35 (1.6525) | 121.40 (1.6525)
  Standing Diastolic BP: 4 hour post Maraviroc dose | 77.29 (1.0102) | 78.38 (1.0102)
  Standing Systolic BP: 6 hour post Maraviroc dose | 118.29 (1.6525) | 120.59 (1.6525)
  Standing Diastolic BP: 6 hour post Maraviroc dose | 73.34 (1.0102) | 76.77 (1.0102)
  Standing Systolic BP: 8 hour post Maraviroc dose | 120.43 (1.6525) | 123.90 (1.6525)
  Standing Diastolic BP: 8 hour post Maraviroc dose | 74.06 (1.0102) | 77.32 (1.0102)
  Standing Systolic BP: 12 hour post Maraviroc dose | 128.38 (1.6525) | 128.65 (1.6525)
  Standing Diastolic BP: 12 hour post Maraviroc dose | 78.65 (1.0102) | 80.91 (1.0102)
Statistical Analysis 1: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 1.5 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; Sequence, period, time, treatment, & time by treatment interaction as fixed effects, subject within sequence as random effect. Baseline was covariate; Mean Difference (Final Values) = -1.11, 90% CI [-3.80 to 1.59]
Statistical Analysis 2: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 1.5 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.93, 90% CI [-3.55 to -0.31]
Statistical Analysis 3: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.99, 90% CI [-7.69 to -2.30]
Statistical Analysis 4: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.96, 90% CI [-4.58 to -1.34]
Statistical Analysis 5: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2.5 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.88, 90% CI [-7.58 to -2.19]
Statistical Analysis 6: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2.5 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.82, 90% CI [-5.44 to -2.20]
Statistical Analysis 7: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 3 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.05, 90% CI [-4.74 to 0.64]
Statistical Analysis 8: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 3 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.76, 90% CI [-3.38 to -0.15]
Statistical Analysis 9: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 4 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.08, 90% CI [-4.77 to 0.62]
Statistical Analysis 10: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 4 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.88, 90% CI [-2.49 to 0.74]
Statistical Analysis 11: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 6 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.30, 90% CI [-4.99 to 0.39]
Statistical Analysis 12: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 6 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.85, 90% CI [-2.47 to 0.77]
Statistical Analysis 13: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 8 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.22, 90% CI [-6.91 to -1.52]
Statistical Analysis 14: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 8 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.51, 90% CI [-4.13 to -0.90]
Statistical Analysis 15: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 12 hour post-dose for supine systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.94, 90% CI [-4.63 to 0.76]
Statistical Analysis 16: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 12 hour post-dose for supine diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.32, 90% CI [-3.94 to -0.70]
Statistical Analysis 17: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 1.5 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.36, 90% CI [-8.22 to -0.50]
Statistical Analysis 18: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 1.5 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.93, 90% CI [-6.29 to -1.56]
Statistical Analysis 19: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.91, 90% CI [-10.77 to -3.05]
Statistical Analysis 20: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.79, 90% CI [-8.15 to -3.42]
Statistical Analysis 21: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2.5 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.80, 90% CI [-9.66 to -1.94]
Statistical Analysis 22: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2.5 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.65, 90% CI [-9.01 to -4.29]
Statistical Analysis 23: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 3 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.27, 90% CI [-8.13 to -0.41]
Statistical Analysis 24: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 3 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.65, 90% CI [-6.01 to -1.29]
Statistical Analysis 25: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 4 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.05, 90% CI [-5.91 to 1.81]
Statistical Analysis 26: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 4 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.09, 90% CI [-3.46 to 1.27]
Statistical Analysis 27: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 6 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.30, 90% CI [-6.16 to 1.56]
Statistical Analysis 28: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 6 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.43, 90% CI [-5.79 to -1.06]
Statistical Analysis 29: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 8 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.47, 90% CI [-7.33 to 0.39]
Statistical Analysis 30: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 8 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.26, 90% CI [-5.62 to -0.90]
Statistical Analysis 31: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 12 hour post-dose for standing systolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.27, 90% CI [-4.13 to 3.59]
Statistical Analysis 32: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 12 hour post-dose for standing diastolic BP Vardenafil minus Placebo A total sample size of 18 subjects provides 90% confidence intervals for the difference between vardenafil and placebo of ±5.90 on the standing diastolic BP with 98% coverage probability at each time postdose; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.26, 90% CI [-4.62 to 0.10]

2. Secondary Outcome: Standing and Supine Pulse Rate
Description: Supine pulse rate measurement was taken after subject rested for 5 minutes supine. Subject sat for 2 minutes, then stood for 2 minutes and standing measurement taken. Duplicate supine and standing pulse rate measurements taken per protocol. Average of duplicate measurements calculated prior to data analysis.
Time Frame: 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours post Vardenafil or Placebo dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Maraviroc + Vardenafil (Treatment A) | Maraviroc + Placebo (Treatment B)
Number analyzed (Participants) | 18 | 18
beats per minute (bpm)
  Supine pulse rate: 1.5 hours post Maraviroc dose | 67.56 (1.3482) | 60.61 (1.3482)
  Supine pulse rate: 2 hours post Maraviroc dose | 66.20 (1.3482) | 60.69 (1.3482)
  Supine pulse rate: 2.5 hours post Maraviroc dose | 61.64 (1.3482) | 58.00 (1.3482)
  Supine pulse rate: 3 hours post Maraviroc dose | 60.42 (1.3482) | 57.53 (1.3482)
  Supine pulse rate: 4 hours post Maraviroc dose | 60.22 (1.3482) | 58.16 (1.3482)
  Supine pulse rate: 6 hours post Maraviroc dose | 71.39 (1.3482) | 65.94 (1.3482)
  Supine pulse rate: 8 hours post Maraviroc dose | 67.67 (1.3482) | 63.55 (1.3482)
  Supine pulse rate: 12 hours post Maraviroc dose | 71.25 (1.3482) | 67.80 (1.3482)
  Standing pulse rate: 1.5 hours post Maraviroc dose | 85.78 (1.6885) | 78.45 (1.6885)
  Standing pulse rate: 2 hours post Maraviroc dose | 85.16 (1.6885) | 78.34 (1.6885)
  Standing pulse rate: 2.5 hours post Maraviroc dose | 82.25 (1.6885) | 77.22 (1.6885)
  Standing pulse rate: 3 hours post Maraviroc dose | 80.05 (1.6885) | 75.34 (1.6885)
  Standing pulse rate: 4 hours post Maraviroc dose | 79.97 (1.6885) | 75.92 (1.6885)
  Standing pulse rate: 6 hours post Maraviroc dose | 93.53 (1.6885) | 87.17 (1.6885)
  Standing pulse rate: 8 hours post Maraviroc dose | 84.41 (1.6885) | 79.34 (1.6885)
  Standing pulse rate: 12 hours post Maraviroc dose | 82.47 (1.6885) | 80.59 (1.6885)
Statistical Analysis 1: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 1.5 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.95, 90% CI [4.18 to 9.72]
Statistical Analysis 2: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.51, 90% CI [2.73 to 8.28]
Statistical Analysis 3: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2.5 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.64, 90% CI [0.87 to 6.42]
Statistical Analysis 4: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 3 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.89, 90% CI [0.12 to 5.67]
Statistical Analysis 5: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 4 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.06, 90% CI [-0.71 to 4.83]
Statistical Analysis 6: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 6 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.45, 90% CI [2.68 to 8.22]
Statistical Analysis 7: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 8 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.12, 90% CI [1.34 to 6.89]
Statistical Analysis 8: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 12 hour post-dose for supine pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.45, 90% CI [0.68 to 6.22]
Statistical Analysis 9: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 1.5 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.33, 90% CI [3.70 to 10.95]
Statistical Analysis 10: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.83, 90% CI [3.20 to 10.45]
Statistical Analysis 11: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 2.5 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.02, 90% CI [1.40 to 8.65]
Statistical Analysis 12: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 3 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.72, 90% CI [1.09 to 8.34]
Statistical Analysis 13: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 4 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.05, 90% CI [0.43 to 7.67]
Statistical Analysis 14: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 6 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.36, 90% CI [2.73 to 9.98]
Statistical Analysis 15: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 8 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.08, 90% CI [1.45 to 8.70]
Statistical Analysis 16: Comparison: Maraviroc + Vardenafil (Treatment A) vs Maraviroc + Placebo (Treatment B); 12 hour post-dose for standing pulse rate Vardenafil minus Placebo; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.88, 90% CI [-1.74 to 5.51]

3. Secondary Outcome: Postural Changes in Systolic and Diastolic Blood Pressure
Description: Postural change calculated as position 1 (standing) value minus the position 2 (supine) value. Baseline was the average of 3 predose measurements at each period. Means of replicates were used in calculations.
Time Frame: Baseline, 6 and 12 hours post dose on Day 1 from the First Day of each Treatment Leg
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Maraviroc + Vardenafil (Treatment A) | Maraviroc + Placebo (Treatment B)
Number analyzed (Participants) | 18 | 18
mm Hg
  Systolic Blood Pressure: Baseline | 3.5 (5.01) | 2.6 (4.34)
  Diastolic Blood Pressure: Baseline | 8.9 (4.69) | 7.5 (3.41)
  Systolic Blood Pressure: 6 hours | 2.2 (5.96) | 1.5 (5.14)
  Diastolic Blood Pressure: 6 hours | 8.4 (4.71) | 9.6 (4.36)
  Systolic Blood Pressure: 12 hours | 5.9 (6.21) | 3.5 (5.69)
  Diastolic Blood Pressure: 12 hours | 11.4 (4.66) | 9.9 (4.18)

4. Secondary Outcome: Postural Changes in Pulse Rate
Description: Postural change calculated as position 1 (standing) value minus position 2 (supine) value. Baseline was the average of the 3 predose measurements at each period. Means of Replicates were used in calculations.
Time Frame: Baseline, 6 and 12 hours post dose on Day 1 from the First Day of each Treatment Leg
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Maraviroc + Vardenafil (Treatment A) | Maraviroc + Placebo (Treatment B)
Number analyzed (Participants) | 18 | 18
beats per minute (bpm)
  Baseline | 16.0 (7.32) | 14.3 (8.05)
  6 hours | 22.9 (9.10) | 20.4 (8.25)
  12 hours | 12.0 (6.85) | 12.0 (8.60)

5. Secondary Outcome: Number of Subjects With Postural Hypotension
Description: Postural (orthostatic) hypotension defined as 1) decrease in standing-supine diastolic blood pressure (BP) greater than or equal to 10 mm Hg; 2) decrease in standing-supine systolic BP greater than or equal to 20 mm Hg; or 3) standing systolic BP less than 90 mm Hg. Assessed at Period 1 and Period 2 BP measurement timepoints post maraviroc dose.
Time Frame: Period 1 and Period 2 (up to 8 days)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Maraviroc + Vardenafil (Treatment A) | Maraviroc + Placebo (Treatment B)
Number analyzed (Participants) | 18 | 18
participants | 0 | 0

ADVERSE EVENTS:
Groups:
- Maraviroc Run-In: All subjects received 3 to 4 days of maraviroc 300 mg twice daily (BID) before receiving single oral doses of either vardenafil 20 mg (Treatment A) or placebo (Treatment B).
- Maraviroc + Vardenafil (Treatment A): On Days 1 through 3 during Period 1, and Days 1 through 2 during Period 2, a maraviroc 300 mg tablet was to be taken orally BID to achieve steady state. On Day 4 of Period 1, and Day 3 of Period 2, a single dose of vardenafil 20 mg tablet was administered orally 1 hour post maraviroc dosing.
- Maraviroc + Placebo (Treatment B): On Days 1 through 3 during Period 1, and Days 1 through 2 during Period 2, a maraviroc 300 mg tablet was taken orally BID to achieve steady state. On Day 4 of Period 1, and Day 3 of Period 2, a single dose of non-matching placebo tablet was administered orally 1 hour post maraviroc dosing.
Arm/Group | Maraviroc Run-In | Maraviroc + Vardenafil (Treatment A) | Maraviroc + Placebo (Treatment B)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4 | 16 | 5
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Maraviroc Run-In | Maraviroc + Vardenafil (Treatment A) | Maraviroc + Placebo (Treatment B)
Headache (Nervous system disorders) | 1/18 | 8/18 | 1/18
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/18 | 8/18 | 0/18
Hot flush (Vascular disorders) | 0/18 | 8/18 | 0/18
Erection increased (Reproductive system and breast disorders) | 0/18 | 3/18 | 0/18
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0/18 | 2/18 | 1/18
Dizziness (Nervous system disorders) | 0/18 | 2/18 | 2/18
Fatigue (General disorders) | 0/18 | 2/18 | 0/18
Abdominal discomfort (Gastrointestinal disorders) | 1/18 | 1/18 | 0/18
Diarrhoea (Gastrointestinal disorders) | 0/18 | 1/18 | 0/18
Phosphenes (Eye disorders) | 0/18 | 1/18 | 0/18
Nausea (Gastrointestinal disorders) | 0/18 | 1/18 | 0/18
Suprapubic pain (General disorders) | 1/18 | 1/18 | 0/18
Somnolence (Nervous system disorders) | 0/18 | 1/18 | 0/18
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0/18 | 1/18 | 0/18
Rash (Skin and subcutaneous tissue disorders) | 0/18 | 1/18 | 0/18
Tooth fracture (Injury, poisoning and procedural complications) | 1/18 | 1/18 | 1/18
Back pain (Musculoskeletal and connective tissue disorders) | 1/18 | 1/18 | 1/18
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/18 | 1/18 | 1/18
Eye pain (Eye disorders) | 0/18 | 0/18 | 1/18
Dyspepsia (Gastrointestinal disorders) | 0/18 | 0/18 | 1/18
Hepatic enzyme increased (Investigations) | 0/18 | 0/18 | 1/18
Myalgia (Musculoskeletal and connective tissue disorders) | 0/18 | 0/18 | 1/18
Dizziness postural (Nervous system disorders) | 0/18 | 0/18 | 1/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.